CLINICAL TRIAL: NCT03386955
Title: An Open-label, Single Arm, Phase I/IIa Study to Evaluate Safety, Dose Escalation Tolerability, Pharmacokinetics and Antineoplastic Activity of the BPI-7711 Capsule in Patients With EGFR Mutation Advanced or Recurrent NSCLC
Brief Title: BPI-7711 Capsule in Patients With EGFR Mutation T790M Positive Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beta Pharma Shanghai (Industry)
Responsible Party: Sponsor
Organization: Beta Pharma, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPI-7711-2015-001
Record Dates: First submitted 2017-11-04; First posted 2017-12-29 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — rezivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BPI-7711 treatment (Experimental): Phase I: Patients in dose escalation group will receive single dose of BPI-7711 on day -7 and start receive the 21 days/cycle continuous treatment once a day after 7 day washout period. Patients in the extension group will receive BPI-7711 once a day with the selected doses.
  Phase IIa: Patients will receive BPI-7711 capsule(recommend phase 2 dose) as the first line treatment.
  Interventions: Drug: BPI-7711 Capsule

INTERVENTIONS:
Drug: BPI-7711 Capsule — Phase I: BPI-7711 capsule(30mg, 60mg, 120mg, 180mg, 240mg...) Phase IIa: BPI-7711 capsule(with recommend phase II dose)
  Other Names: BPI-7711; BPI7711 Capsule

SUMMARY:
Lung cancer has the highest incidence rate in China and is also a very common cancer in the world. BPI-7711 is a new drug developed for patients with non-small cell lung cancer.

The purpose of this study is to evaluate the safety, efficacy and PK profile of BPI-7711. The first part of the study will recruit 3~6 patients for different dose levels to evaluate safety. The dose will increase from the lowest level. The second part of the study is the dose expansion. Once efficacy is observed in the dose increasing process, additional 20~30 patients will be enrolled to further evaluate the anti-tumor efficacy. A recommended dose will be selected for Phase II study.

DETAILED DESCRIPTION:
This is a single arm, open label study, including phase I (a "dose escalation" part and a "dose extension" part) and phase IIa.

Dose escalation: on the basis of the traditional "3+3" dose escalation plan; single dose PK test is added. The subjects of each dose group will first be given a single dose, and blood samples be collected for PK analysis. 7 days (wash-out period) after single dose delivery, an additional 21 days of continuous multiple dose delivery will be given as a treatment cycle to evaluate the dose limiting toxicity (DLT). The initial dose will be 30 mg once a day. In the initial dose group, the second subject will be enrolled and administered with the study drug 7 days after the first dosing (single dose) to the first subject. If there is no occurrence of serious or unexplainable safety event, the subsequent following-up subjects will be enrolled and receive the dose. If suspected safety event occurs, the investigator will discuss with the sponsor whether to delay dose delivery to the following-up subjects of the said group.

Every dose escalation group will enroll 3 to 6 subjects. Dose adjustment will be based on the following scheme:

* If there is 0 case of DLT in 3 subjects of the initial dose group in the first treatment cycle, then the treatment dose of the subsequent 3 patients will be increased to level 2.
* If there is 1 case of DLT in 3 subjects of the initial dose group in the first treatment cycle, then additional 3 patients will be enrolled in the group and accept the level 1 dose treatment.

  * If there is 0 case of DLT in the 3 new subjects, the dose will be increased to level 2.
  * If there is ≥1 case of DLT in the 3 new subjects, the principal investigator and the sponsor will discuss to determine the next step dose scheme.
* If there are ≥2 cases of DLT in 3 subjects of the initial dose group, the principal investigator and the sponsor will meet to discuss the alternative dose delivery scheme.

The same dose escalation rules shall be applicable to the following dose groups. Based on available tolerance, safety, and PK data, recommended Phase II dose (RP2D) will be selected.

Dose extension group: If a certain dose is found to be safe and effective, dose expansion will be initiated and about 20-30 subjects will be enrolled into that dose level. There will be no DLT evaluation for subjects of the dose extension study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects signs and dates the informed consent form before receiving any treatment or test sample collection related to the study.
* Male or female, ≥18 and ≤75 years of age when signing the informed consent.
* Locally advanced or metastatic non-small cell lung cancer (NSCLC) verified by histology or cytology, and no longer suitable for radical surgery or radiation therapy.
* ECOG scoring (PS) of physical conditions 0-1, and there is no deterioration 2 weeks before enrolled to the study. The expected survival is not less than 12 weeks.
* Phase I: Disease progressed after EGFR-TKI treatment as proved by radiological evidence. For dose level which does not provide satisfying efficacy in the escalation group, patients must receive chemo therapy before enrolled into that dose, unless not suitable for chemotherapy judged by investigator. Patients must have documented radiological progression before enrolled into the study. Phase IIa: Patients must be treatment- naïve for locally advanced or metastatic NSCLC. Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy, investigational agents) provided all other entry criteria are satisfied
* At least 1 measurable lesion based on the RECIST1.1 criteria. If the subject has only 1 measurable lesion, the baseline CT must be performed before biospy or at least 14 days after biopsy. The lesion received radiotherapy does not count as measurable lesion or a biopsy lesion unless it shows obvious progression after radiotherapy. Brain metastases and irradiated lesions are not taken as target lesions.
* Prior to enrollment, a central laboratory testing report confirmed the tumor has EGFR positive gene mutation sensitive to EGFR-TKI treatment (including G719X, exon 19 loss, L858R, L861Q etc.).
* Phase I: Central lab tissue tests confirm T790M positive for the biopsy, plasma, or cytology samples collected after imaging examination with clear disease progression post last treatment. Subject should provide formalin fixed and paraffin embedded tumor tissue block or 5 pieces of 4-5µm thick undyed slices, or should agree to do tumor tissue biopsy.
* The clinical laboratory examination results shall meet the following criteria:

  1. Blood platelet ≥100×10^9/L
  2. Absolute neutrophil counting（ANC）≥1.5×10^9/L
  3. Hemoglobin（Hgb）≥90 g/L
  4. Total bilirubin (TBil) ≤1.5 times of upper normal limit（ULN） (≤3 times of ULN is allowed if there is liver metastasis)
  5. Alanine aminotransferase (ALT) and aspertate aminotransferase (AST) ≤3 times of ULN (≤5 times of ULN is allowed if there is liver metastasis)
  6. Creatinine ≤1.5times of ULN or creatinine clearance≥50 mL/min.
  7. Mean resting corrected QT interval (QTc) ≤470 msec obtained from 3 electrocardiograms (ECGs).
  8. If the subject is not taking anticoagulants, the International Standardization Ratio (INR) ≤1.5 and APTT ≤1.5 times of ULN. For patients who are being treated with heparin anticoagulant therapy, if these indicators have no abnormality, and then they can be enrolled. For subjects who are receiving warfarin anticoagulant therapy, within 28 days before enrolled into the study, relating to INR, use stable dose warfarin.
* Able to swallow the study drug.
* Female subjects should take effective contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential.
* Male patient subjects are willing to use barrier contraception.
* Except hair loss and stable below level 2 peripheral nerve toxicity, any clinical toxicity related to previous treatment before enrollment must restore to pre-treatment or level 1.

Exclusion Criteria:

* Anti-cancer treatment with first/second generation of EGFR-TKI (e.g., Icotinib, gefitinib, erlotinib afatinib, dacomitinib, etc) within 8 days (approximately 5 times of half-life) before first dosing in the study.
* Received treatment targeted for T790M positive mutation, or participated in clinical trials for such types of drugs, e.g., AZD9291, CO-1686 and other third-generation TKI therapy.
* Any cytotoxic chemotherapy, investigational agents or anticancer drugs for the treatment of advanced NSCLC from a previous treatment regimen or clinical study within 14 days prior to the first dose of study treatment.
* Any of the following cardiac criteria: resting corrected QT interval (QTcF) > 470 msec; Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, III-degree heart block, II-degree heart block, PR interval >250 msec; Factors that may increase the risk of QTc prolongation or risk of arrhythmic events such as symptomatic heart failure - New York Heart Association (NYHA) Class II-IV, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT intervals.
* Past interstitial lung disease, drug induced interstitial lung disease, radiation pneumonia that needs steroid therapy, or any evidence of clinically. active interstitial lung disease.
* The known active infection, such as hepatitis B, hepatitis C and human immunodeficiency virus (HIV) infection. Patients with well-controlled hepatitis B can be enrolled to the study, and can receive antiviral treatment.
* Patients with other malignant tumor and still under treatment, or have recurrent or associated other malignant tumor within the last 5 years are not eligible. Cervical cancer in situ eradication therapy, non-melanoma skin cancer, superficial bladder tumor (noninvasive tumor), or carcinoma in situ with no recurrence, nor relevant treatment in 3 years after eradication treatment, may be eligible.
* Judged by investigators, clear digestive tract disorder which may interfere with BPI-7711 absorption (for example, obvious uncontrolled inflammatory gastrointestinal diseases, abdominal colostomy within 6 months or past history of gastrointestinal perforation, intestinal wide excision and the need for tube feeding or parenteral fluids/nutrition supplementation).
* Spinal cord compression, metastases of the meninges, and brain metastases with obvious symptoms. cannot be enrolled. The following cases of brain metastases without symptoms can be enrolled: Brain metastases without obvious symptoms diagnosed at screening visit, steroids and/or local treatment not required judged by investigator; Brain metastases without obvious symptoms after local treatment (such as radiotherapy), and steroids and/or antiepileptic therapy has stopped for at least 7 days before the first dosing of study drug.
* Local radiotherapy to alleviate the disease within 1 week before first dosing of the study drug; more than 30% bone marrow radiotherapy or with a wide field of radiotherapy within 4 weeks before first dosing of the study drug.
* ≤4 weeks before major surgery or ≤2 weeks before minor surgery before the first day of administration of the study drug.
* Any unstable factor or factors that may endanger the safety of the patients or affect the subjects' compliance to procedures and requirements of this study.
* Leukocyte-depleted whole blood transfusion within the 120 days before collecting genetic testing samples.
* Pregnant or breast-feeding women.
* All subjects must have enough mental behavior ability, understand the nature and significance of the study, as well as the risks associated with this study.
* Drug abuse, alcoholic addiction, medical and mental illness and social barriers which may interfere the subjects' participation in the study or affect study result evaluation judged by investigator. Any factor that the investigator believes may make the candidates not suitable to receive study drug. The candidates are unwilling or unable to comply with the requirements of the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity ( DLT). | From first dosing ( Day -7) to the last dosing of Cycle 1 ( Day 28).
  DLT to be evaluated according to NCI CTCAE V4.03

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of BPI-7711 and its main metabolites. | Pre-dose, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 48h, 72h, 120h, 144h post first dose on Day -7.
  Collect and analyze the blood concentration data of BPI-7711 and its main metabolites on Day-7~Day-1 at designated time points.
Peak Plasma Time (tmax) of BPI-7711 and its main metabolites after single dose. | Pre-dose, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 48h, 72h, 120h, 144h post first dose on Day -7.
  Collect and analyze the blood concentration data of BPI-7711 and its main metabolites on Day-7~Day-1 at designated time points.
Area under the plasma concentration versus time curve (AUC) of BPI-7711 and its main metabolites after single dose. | Pre-dose, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 48h, 72h, 120h, 144h post first dose on Day -7.
  Collect and analyze the blood concentration data of BPI-7711 and its main metabolites on Day-7~Day-1 at designated time points.
Clearance of BPI-7711 and its main metabolites after single dose. | Pre-dose, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 48h, 72h, 120h, 144h post first dose on Day -7.
  Collect and analyze the blood concentration data of BPI-7711 and its main metabolites on Day-7~Day-1 at designated time points.
Half life of BPI-7711 and its main metabolites after single dose. | Pre-dose, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h, 48h, 72h, 120h, 144h post first dose on Day -7.
  Collect and analyze the blood concentration data of BPI-7711 and its main metabolites on Day-7~Day-1 at designated time points.
Blood concentration of BPI-7711 and its main metabolites after single dose under steady state. | Pre-dose of Cycle1 Day1, 8, 15. Pre-dose, 1h, 1.5h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 24h post dose on Cycle 2 Day1
  Collect and analyze the blood concentration data of BPI-7711 and its main metabolites on Cycle 1 Day1, Cycle Day 8, Cycle 1 Day 15 and Cycle 2 Day1 at designated time. points.
Objective response rate (ORR) of BPI-7711 capsule. | At screening, and every two cycles from the first multiple dose on Cycle 1 Day 1( 21 days as one cycle) until the date of first documented progression, death or withdrawal from study, whichever came first, assessed up to 20 months.
  Objective response rate evaluated by CT, MRI examination results according to RECIST 1.1.
Best objective response (BOR) of BPI-7711 capsule. | At screening, and every two cycles from the first multiple dose on Cycle 1 Day 1( 21 days as one cycle) until the date of first documented progression, death or withdrawal from study, whichever came first, assessed up to 20 months.
  Best objective response evaluated by CT, MRI examination results according to RECIST 1.1.
Disease control rate ( DCR) of BPI-7711 capsule. | At screening, and every two cycles from the first multiple dose on Cycle 1 Day 1( 21 days as one cycle) until the date of first documented progression, death or withdrawal from study, whichever came first, assessed up to 20 months.
  Disease control rate evaluated by CT, MRI examination results according to RECIST 1.1.
Duration of response ( DoR) of BPI-7711 capsule. | At screening, and every two cycles from the first multiple dose on Cycle 1 Day 1( 21 days as one cycle) until the date of first documented progression, death or withdrawal from study, whichever came first, assessed up to 20 months.
  Duration of response evaluated by CT, MRI examination results according to RECIST 1.1.
Progression free survival (PFS) of BPI-7711 capsule. | At screening, and every two cycles from the first multiple dose on Cycle 1 Day 1( 21 days as one cycle) until the date of first documented progression, death or withdrawal from study, whichever came first, assessed up to 20 months.
  Progression free survival evaluated by CT, MRI examination results according to RECIST 1.1.

OTHER OUTCOMES:
EGFR mutation testing. | At screening and every two cycles( 21 days as a cycle) from Cycle 1 Day1 until the date of first documented progression, death or withdrawal from study, whichever came first, assessed up to 20 months.
  To test EGFR mutation in plasma circulating tumor DNA (ctDNA).
T790M mutation testing. | At screening and every two cycles( 21 days as a cycle) from Cycle 1 Day1 until the date of first documented progression, death or withdrawal from study, whichever came first, assessed up to 20 months.
  To test T790M mutation in plasma circulating tumor DNA (ctDNA).

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang S, Wu S, Zhao Y, Chen G, Zhu B, Li X, Wang K, Shi J, Cang S, Yao W, Fan Y, Fang J, Zhang L, Zhou J, Wu L, Zheng R, Huang M, Pan Y, Yang Z, Sun M, Yu H, Wang D, Huang J, Wang L, Shu Y, Chen Z, Liu C, Li J, Liu J, Sun S, Guo Y, Meng Z, Liu Z, Han Z, Wu G, Lu H, Ma R, Hu S, Zhao G, Zhang L, Liu Z, Xie C, Zhong D, Zhao H, Bi M, Yi S, Guo S, Yi T, Li W, Lin Y, Chen Z, Zhuang Z, Guo Z, Greco M, Wang T, Zhou A, Shi Y. Central nervous system efficacy of rezivertinib (BPI-7711) in advanced NSCLC patients with EGFR T790M mutation: A pooled analysis of two clinical studies. Lung Cancer. 2023 Jun;180:107194. doi: 10.1016/j.lungcan.2023.107194. Epub 2023 Apr 17. PMID 37163774
- [Derived] Shi Y, Zhou J, Zhao Y, Zhu B, Zhang L, Li X, Fang J, Shi J, Zhuang Z, Yang S, Wang D, Yu H, Zhang L, Zheng R, Greco M, Wang T. Results of the phase IIa study to evaluate the efficacy and safety of rezivertinib (BPI-7711) for the first-line treatment of locally advanced or metastatic/recurrent NSCLC patients with EGFR mutation from a phase I/IIa study. BMC Med. 2023 Jan 8;21(1):11. doi: 10.1186/s12916-022-02692-8. PMID 36617560
- [Derived] Shi Y, Zhao Y, Yang S, Zhou J, Zhang L, Chen G, Fang J, Zhu B, Li X, Shu Y, Shi J, Zheng R, Wang D, Yu H, Huang J, Zhuang Z, Wu G, Zhang L, Guo Z, Greco M, Li X, Zhang Y. Safety, Efficacy, and Pharmacokinetics of Rezivertinib (BPI-7711) in Patients With Advanced NSCLC With EGFR T790M Mutation: A Phase 1 Dose-Escalation and Dose-Expansion Study. J Thorac Oncol. 2022 May;17(5):708-717. doi: 10.1016/j.jtho.2022.01.015. Epub 2022 Feb 15. PMID 35181498